CLINICAL TRIAL: NCT06270966
Title: Cognitive Remediation Virtual Reality Tool a Recovery-oriented Project for People With Mild Cognitive Impairment: a Feasibility Randomized Clinical Trial
Brief Title: Cognitive Remediation VR Tool for People With MCI: a Feasibility RCT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Cagliari (Other)
Responsible Party: Principal Investigator, Mauro Giovanni Carta, Principal Investigator, University of Cagliari
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 28287 08/11/2023
Record Dates: First submitted 2024-02-13; First posted 2024-02-21 (Actual); Last update posted 2024-02-21 (Actual); Status verified 2024-02

CONDITIONS: Mild Cognitive Impairment; Cognitive Remediation; Virtual Reality; Psychiatric Rehabilitation
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual Reality Cognitive Remediation + treatment as usual (Experimental): 15 Participants with more than 65 years and with MCI diagnosis will undergo a cognitive remediation program using fully immersive VR. Participants will continue with standard care during the experimental intervention
  Interventions: Device: Virtual Reality Cognitive Remediation
- Treatment as usual (No Intervention): The control group, 15 participants with more than 65 years and with MCI diagnosis, will continue with standard care.

INTERVENTIONS:
Device: Virtual Reality Cognitive Remediation — Participants will undergo a 3-months cognitive remediation program using fully immersive VR with two sessions per week. Each session will last a maximum of sixty minutes and will be supervised by expert health professionals. The experimental group participated in an immersive VR-based CR program using the "CEREBRUM" software designed by clinicians and experts specializing in cognitive rehabilitation.
  CEREBRUM provides 52 exercises: Attention, Working Memory, Memory and Learning and Cognitive Estimates. The intervention included 24 sessions.
  Arms: Virtual Reality Cognitive Remediation + treatment as usual

SUMMARY:
The need to promote research in active aging trough multidisciplinary and innovative approaches is strongly indicated by the European Union. Our study aims to assess the feasibility and provide a preliminary measure of effectiveness for an intervention using immersive virtual reality (VR) technology for cognitive remediation (CR) in individuals with Mild Cognitive Impairment (MCI)

DETAILED DESCRIPTION:
The European Union emphasizes the need to promote research in active aging trough multidisciplinary and innovative approaches, addressing challenges related to neurodegenerative diseases in old adults. Our study aims to assess the feasibility and provide a preliminary measure of effectiveness for an intervention using immersive virtual reality (VR) technology for cognitive remediation (CR) in individuals with Mild Cognitive Impairment (MCI).

Methods: A feasibility randomized controlled clinical trial will involve 30 individuals who are over 65 years old, both sex, who have received the diagnosis of MCI, randomly assigned to experimental condition or control group. Both groups will continue to receive standard pharmacological therapy (TAU). The experimental group will undergo a 3-months cognitive remediation program with fully immersive VR with two sessions per week (each session of sixty minutes). The control group will continue with TAU.

Feasibility will be assessed based on tolerability, including dropout rates and acceptability, (proportion of recruited participants among those considered eligible) and side effects. The preliminary measures of effectiveness will be evaluated on cognitive functions, quality of life, biological and social rhythms, anxiety and depressive.

ELIGIBILITY:
Inclusion Criteria:

* age 65 and above, a diagnosis of MCI based on DSM-IV criteria [American Psychiatric Association, 2000]

Exclusion Criteria:

* failure to meet inclusion criteria, a diagnosis of epilepsy or severe visual impairments due to potential risks associated with extensive virtual reality stimulation, and severe illnesses impeding bi-weekly intervention attendance

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-03-07 (Estimated); Primary Completion 2024-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Side effects; Dropout rates; Proportion of recruited participants among those considered eligible | T0 (0 weeks); T1 (12 weeks)
  Feasibility will be assessed based on tolerability, including dropout rates and acceptability, which considers the proportion of recruited participants among those considered eligible and side effects.

SECONDARY OUTCOMES:
Short Form Health Survey, 12 items (SF-12) | T0 (0 weeks); T1 (12 weeks); T2 (36 weeks); (72 weeks)
  Preliminary measures of effectiveness on quality of life, 12 items
Brief Social Rhythms Scale (BSRS) | T0 (0 weeks); T1 (12 weeks); T2 (36 weeks); (72 weeks)
  Preliminary measures of effectiveness on biological and social rhythms, 10 items
Patient Health Questionnaire (PHQ-9) | T0 (0 weeks); T1 (12 weeks); T2 (36 weeks); (72 weeks)
  Preliminary measures of effectiveness on depressive symptoms, 9 Items
Generalized Anxiety Disorder-7 item (GAD-7) | T0 (0 weeks); T1 (12 weeks); T2 (36 weeks); (72 weeks)
  Preliminary measures of effectiveness on anxiety, 7 items
Addenbrooke's Cognitive Examination (ACE-R) | T0 (0 weeks); T1 (12 weeks); T2 (36 weeks); (72 weeks)
  Preliminary measures of effectiveness on general cognitive functions, the neuropsychological tests is used to identify cognitive impairment in conditions such as dementia.
Matrix test | T0 (0 weeks); T1 (12 weeks); T2 (36 weeks); (72 weeks)
  Preliminary measures of effectiveness on attention
Rey's Word Test | T0 (0 weeks); T1 (12 weeks); T2 (36 weeks); (72 weeks)
  Preliminary measures of effectiveness on memory
Trail Making Test (TMT) | T0 (0 weeks); T1 (12 weeks); T2 (36 weeks); (72 weeks)
  Preliminary measures of effectiveness on executive function
Digit Span | T0 (0 weeks); T1 (12 weeks); T2 (36 weeks); (72 weeks)
  Preliminary measures of effectiveness on memory
Stroop Test | T0 (0 weeks); T1 (12 weeks); T2 (36 weeks); (72 weeks)
  Preliminary measures of effectiveness on executive function
Frontal Assessment Battery (FAB) | T0 (0 weeks); T1 (12 weeks); T2 (36 weeks); (72 weeks)
  Preliminary measures of effectiveness on executive function
Cognitive Estimates Test (CET) | T0 (0 weeks); T1 (12 weeks); T2 (36 weeks); (72 weeks)
  Preliminary measures of effectiveness on executive function
Rey Figure Test | T0 (0 weeks); T1 (12 weeks); T2 (36 weeks); (72 weeks)
  Preliminary measures of effectiveness on visual spatial function

CONTACTS AND LOCATIONS:
Locations (1):
- San Giovanni di Dio Hospital, Cagliari, CA, Italy